CLINICAL TRIAL: NCT00152048
Title: A 24 Week Randomised Double Blind Placebo Controlled Study to Evaluate the Atrophogenic Potential of Eflornithine in the Treatment of Women With Excessive Facial Hair
Brief Title: Evaluation of Eflornithine on Facial and Forearm Skin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SPD488-401; 2004-000726-78 (EudraCT Number)
Record Dates: First submitted 2005-09-08; First posted 2005-09-09 (Estimated); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Hirsutism
MeSH Terms: conditions — Hirsutism | interventions — Eflornithine

INTERVENTIONS:
Drug: Eflornithine hydrochloride

SUMMARY:
The purpose of this study is to evaluate whether regular use of eflornithine 11.5% cream in treating women with facial hair will induce skin damage (atrophy) on the face and/or forearms

ELIGIBILITY:
Inclusion Criteria:

* Female subjects with clinical diagnosis of facial hirsutism/excessive facial hair
* Women of childbearing potential must agree to use an effective form of birth control for the duration of the study
* Skin type I-IV
* Customary frequency of removal of facial hair two or more times per week

Exclusion Criteria:

* Pregnant or lactating women
* Severe inflammatory acne or presence of significant scarring on the face
* History of skin malignancy
* Connective tissue disorders

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78
Dates: Start 2004-11-30 (Actual); Study Completion 2005-10-31 (Actual)

PRIMARY OUTCOMES:
Change in facial skin thickness measured by ultrasound at 24 weeks

SECONDARY OUTCOMES:
Skin biopsies
Histology and histochemistry in the dermis
Physician Global Assessment
Subject Self-Assessment Questionnaire